CLINICAL TRIAL: NCT05506163
Title: Development and Validation of a Predictive Model for Postoperative Pulmonary Complications in Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: PPC20210110
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pulmonary Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training set: The whole cohort is randomly assigned to a training cohort and validation cohort.
- validation set: The whole cohort is randomly assigned to a training cohort and validation cohort.

SUMMARY:
Although several clinical predictive models have been developed to predict postoperative pulmonary complications, few predictive models have been developed for elderly patients. In this study, the researchers aimed to develop a new, simplified model to assess the risk of postoperative pulmonary complications in elderly patients using perioperative database information.

DETAILED DESCRIPTION:
Postoperative pulmonary complications occur frequently, which is an important cause of death and morbidity. Age has always been an significant predictor of postoperative pulmonary complications. With an aging population worldwide, more and more elderly people are undergoing surgery due to the expansion of surgical indications. As a result of this phenomenon, the elderly are also an important group for the prediction and intervention of postoperative pulmonary complications. In order to better assess the risk of postoperative pulmonary complications in elderly patients, we constructed a model using database information.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* receiving invasive ventilation during general anesthesia for surgery

Exclusion Criteria:

* preoperative mechanical ventilation
* operations related to previous postoperative complications
* a second operation after surgery
* organ transplantation
* discharged within 24 hours after surgery
* cardiac and thoracic surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: older patients received general anesthesia in Wuhan Union Hospital from January 1, 2014 to December 31, 2019.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2022-09-22 (Estimated); Study Completion 2022-09-22 (Estimated)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | within one week after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China